CLINICAL TRIAL: NCT03339427
Title: Study of Vitamin D Deficiency on Cardiovascular Disease and the Effect of Vitamin D Supplementation
Brief Title: Intervention Study of Vitamin D Supplementation to Prevent Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chunlin Li, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VitD301
Record Dates: First submitted 2014-06-19; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; cardiovascular; muscle power
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D,capsule (Active Comparator): A total of 150 subjects were recruited in the vitamin D supplementation group.
  Interventions: Other: vitamin D
- control (Other): A total of 150 subjects were recruited in the control group.
  Interventions: Other: control

INTERVENTIONS:
Other: vitamin D — different doses of vitamin D supplementation
  Arms: vitamin D,capsule
Other: control — control group
  Arms: control

SUMMARY:
This is a 9 months, randomized, single center, open-label, parallel-group study to compare the efficacy and safety parameters of vitamin D supplementation in vitamin D deficiency subjects in China.

DETAILED DESCRIPTION:
This is a 9 months, randomized, single center, open-label, parallel-group study to compare the efficacy and safety parameters of vitamin D supplementation in vitamin D deficiency subjects in China.

Eligibility for participation will be determined by medical history, physical examination, and laboratory results obtained during a screening visit. About 300 subjects with vitamin D insufficiency or deficiency will be included in this study. All subjects will be given informed consent before starting any examination and test. The following data of all subject will be collected: liver and kidney function, HbA1c, fasting blood glucose, fasting lipid profile, serum calcium, serum phosphate, parathyroid hormone, 25-hydroxy vitamin D(25OHD), serum procollagen type I N propeptide, serum C-terminal telopeptide of type I collagen, s-CTX and muscle power and balance.

After baseline data are collected, eligible subjects will be randomized into each group at a 1:1 ratio (150 for control group and 150 for vitamin D supplementation group, less than 20% drop-off rate is acceptable for this study). The initial vitamin D doses will be based on 25OHD levels at basis, and this dosage may be changed according be the level of 25OHD until the end of this study.

All subjects in the control group will be followed every half year. All subjects in the vitamin D group will be followed by visiting clinic, and will be titrated their doses. Dose adjustment should be aimed at achieving the following 25OHD targets: 30ng/ml. If above 25OHD target has not been achieved, vitamin D dose should be adjusted. Clinic visit will be conducted 3 months later to collect information, such as serum calcium, 25OHD and adverse events.

Complicated examinations will be repeated again after 9 months treatments for both groups, including physical examination, liver and kidney function, HbA1c, fasting blood glucose, fasting lipid profile, serum calcium, serum phosphate, parathyroid hormone, 25-hydroxy vitamin D(25OHD), serum procollagen type I N propeptide, serum C-terminal telopeptide of type I collagen, s-CTX and muscle power and balance. Data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities. (Trial- related activities are any procedure that would not have been performed during normal management of the subject.)
2. 25OHD<30ng/ml

Exclusion Criteria:

1. Severe systemic disease (including severe heart, liver, kidney and lung diseases, severe infection, mental disorder and connective tissue disease)
2. Primary hyperparathyroidism, other bone disease, malabsorption and other chronic gastrointestinal disease.
3. Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures.
4. Use of systemic or inhaled glucocorticoids or other medication known to interfere with bone metabolism.
5. Use of vitamin D related agents in recent 3 months.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The efficacy on serum 25(OH)VitD level | 9 months
  The change of serum 25(OH)VitD level after vitamin D supplementation
The efficacy on metabolic syndrome | 9 months
  The change of metabolic syndrome after vitamin D supplementation

SECONDARY OUTCOMES:
The efficacy on bone biomarkers | 9 months
  The change of bone biomarkers after vitamin D supplementation
The efficacy on blood pressure | 9 months
  The change of blood pressure after vitamin D supplementation
The efficacy on blood lipid | 9 months
  The change of blood lipid after vitamin D supplementation
The efficacy on blood glucose | 9 months
  The change of blood glucose after vitamin D supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Chunlin Li, M.D&Ph.D, Principal Investigator — PLA General Hospital
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China